CLINICAL TRIAL: NCT04013022
Title: The Effects of Lifelong Endurance and Strength Training on the Central and Peripheral Cardiovascular Responses
Brief Title: Exercise Pressor Reflex and Lifelong Training
Acronym: LEaSTCaRe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Massimo Venturelli, PhD, Assistant Professor, Universita di Verona
Other Study IDs: 30444
Record Dates: First submitted 2019-06-21; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Healthy Aging; Cardiovascular Risk Factor
Keywords: Exercise Pressor Reflex; Metaboreflex; Mechanoreflex; Lifelong exercise training

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Young: Healthy young subjects (age 18 - 30 )
  Interventions: Behavioral: Exercise History
- Old Sedentary: Healthy and sedentary old subjects (age 65 - 75)
  Interventions: Behavioral: Exercise History
- Old Endurance Trained: Healthy old subjects ( age 65 - 75) who participated in endurance sports for ≥30 years, ≥5 hours per week and ≥4 sessions per week
  Interventions: Behavioral: Exercise History
- Old Strength Trained: Healthy old subjects ( age 65 - 75) who participated in resistance training/sports for ≥30 years, ≥5 hours per week and ≥4 sessions per week
  Interventions: Behavioral: Exercise History

INTERVENTIONS:
Behavioral: Exercise History — The groups will be divided based on their exercise history

SUMMARY:
Cardiovascular diseases represent the first mortality cause in the world. Ageing is considered as the most prominent risk factor for this kind of diseases. Also, hypertension represents one of the modifiable risk factors. Blood pressure response to exercise is governed by three systems: central command, baroreflex, and a feedback mechanism originating in the skeletal muscle. An abnormal cardiovascular response to exercise facilitates the occurrence of cardiovascular events. The goal of the study is to characterize the cardiovascular response in lifelong trained individuals and explore the potential benefits of endurance and strength training on cardiovascular regulation to exercise onset.

DETAILED DESCRIPTION:
Population ageing represents a problem both for health outcomes and for social dynamics in the social welfare states. Currently, the over 60 represents the fastest growing segment of the population. Despite a downward trend in the incidence of cardiovascular diseases, they remain the main culprits for what concern mortality rates in the world. Increasing age is considered the major risk factor for cardiovascular mortality.

One of the main components of the cardiovascular response to exercise is dictated by the exercise pressor reflex originating in the exercising muscle and responding to metabolic and mechanical stimuli. Research indicates that at least 20% of the regulation of blood pressure could be ascribed to these cardiovascular reflexes. A dysfunctional reflex-mediated response increases the chances of cardiovascular events that may end up in severe consequences.

Chronic exercise training is recognized to be an important tool to control blood pressure. The mechanisms through which exercise exerts its effect are multiple. Among these, an improvement of the neural control of the reflex originating in the muscle seems a likely contributor. However, at present, the effect of chronic exercise training on the EPR response in the elderly has not been elucidated. The aim of the study is to characterize the central and peripheral cardiovascular response in the lifelong endurance and strength trained elders population.

ELIGIBILITY:
Inclusion Criteria

General:

* Young: 18 - 30, males, non smokers
* Old Sedentary: 65 -75, males, non smokers
* Old Endurance Trained: 65 -75, males, non smokers
* Old Strength Trained: 65 - 75, males, non smokers

Exercise history (different for each group):

* Young: ≤ 5 h/week
* Old Sedentary: ≤ 2h/week
* Old Endurance Trained: ≥ 5 h/week, ≥ 30 years of practice, ≥ 4 sessions/week
* Old Strength Trained: ≥ 5 h/week, ≥ 30 years of practice, ≥ 4 sessions/week

Exclusion Criteria:

* History of cardiovascular events/diseases
* Respiratory, musculoskeletal, renal, and insulin-resistant diseases
* Hypercholesterolemia
* Use of beta-blockers
* BMI ≥ 30

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy population from different age groups and different exercise training history
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-11-29 (Estimated); Study Completion 2021-11-29 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Blood Pressure (MAP) | 1 week after recruitment of the subject - We will measure the changes from baseline to the steady state response ( average of 3rd minute)
  Difference in MAP between groups to post-exercise cuff occlusion
Heart Rate (HR) | 1 week after recruitment of the subject - We will measure the change from baseline to peak (peak response in HR due to PLM)
  Difference in heart rate between groups to passive leg movement (PLM)
Muscle Sympathetic Nerve Activity - Microneurography | 1 week after recruitment - We will measure the change from baseline to mean value (during stimulation)
  Difference in muscle sympathetic nerve activity between groups to the different stimulations

SECONDARY OUTCOMES:
Muscle oxidative capacity in vivo / blood pressure response | 10 days after recruitment - Cross-sectional comparison at one time point only
  Linear regression to check whether an abnormal blood pressure response is explained by the different muscle oxidative capacity measured by NIRS in vivo

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Venturelli, PhD, Principal Investigator — Universita di Verona
Locations (1):
- University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milia R, Roberto S, Mulliri G, Loi A, Marcelli M, Sainas G, Milia N, Marongiu E, Crisafulli A. Effect of aging on hemodynamic response to metaboreflex activation. Eur J Appl Physiol. 2015 Aug;115(8):1693-703. doi: 10.1007/s00421-015-3153-5. Epub 2015 Mar 24. PMID 25802227
- [Background] Groot HJ, Rossman MJ, Garten RS, Wang E, Hoff J, Helgerud J, Richardson RS. The Effect of Physical Activity on Passive Leg Movement-Induced Vasodilation with Age. Med Sci Sports Exerc. 2016 Aug;48(8):1548-57. doi: 10.1249/MSS.0000000000000936. PMID 27031748
- [Background] Boushel R. Muscle metaboreflex control of the circulation during exercise. Acta Physiol (Oxf). 2010 Aug;199(4):367-83. doi: 10.1111/j.1748-1716.2010.02133.x. Epub 2010 Mar 27. PMID 20353495
- [Background] Murphy MN, Mizuno M, Mitchell JH, Smith SA. Cardiovascular regulation by skeletal muscle reflexes in health and disease. Am J Physiol Heart Circ Physiol. 2011 Oct;301(4):H1191-204. doi: 10.1152/ajpheart.00208.2011. Epub 2011 Aug 12. PMID 21841019
- [Background] Markel TA, Daley JC 3rd, Hogeman CS, Herr MD, Khan MH, Gray KS, Kunselman AR, Sinoway LI. Aging and the exercise pressor reflex in humans. Circulation. 2003 Feb 11;107(5):675-8. doi: 10.1161/01.cir.0000055190.81716.ab. PMID 12578866